CLINICAL TRIAL: NCT03648515
Title: Evaluation of the Validity and Reliability of Measurements Made on Intra-oral Images of the Dental Arches Compared to Those Made on Poured Plaster Models in the Assessment of Tooth-size-arch-length-discrepancy, Bolton's Analysis and Little's Index of Irregularity.
Brief Title: Evaluation of the Accuracy of Measurements Made on Images Taken From the Mouth for Dental Arches
Status: Completed | Type: Observational
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Other Study IDs: UDDS-Ortho-11-2018
Record Dates: First submitted 2018-08-24; First posted 2018-08-27 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Malocclusion
Keywords: Validity; Reliability; Reproducibility; Intra-oral images; Plaster models; Digital images; Little's index of irregularity; Bolton's analysis; Tooth-size-arch-length-discrepancy
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Malocclusion patients: Patients with different types of malocclusion will be included. Plaster models will be fabricated after pouring the impressions with hard gypsum.
  Then, digital images of the dental arches of each patient will be taken using a dedicated camera with very high resolution. Finally, digital images of models that were poured with gypsum will be taken also with the same camera and in the same conditions.
  Interventions: Diagnostic Test: Plaster models; Diagnostic Test: Digital Images of the dental arches; Diagnostic Test: Digital images of models

INTERVENTIONS:
Diagnostic Test: Plaster models — The impressions taken of the dental arches will be poured with hard gypsum in order to make use of the models for taking measurements. These measurements will be considered the gold standard.
  Other Names: Study models; Study casts; Poured study models
Diagnostic Test: Digital Images of the dental arches — The dental arches will be captured using a dedicated camera in order to be used for measuring the outcomes.
  Other Names: Intra-oral images
Diagnostic Test: Digital images of models — The poured dental models will be captured using a dedicated camera in order to be used for measuring the outcomes.

SUMMARY:
The general trend in the orthodontic practice is to become digital in many aspects. Since 1980s, digital photographs have been available and they play a principal role in the orthodontic practice for documentation and diagnosis purposes. Now photographs have an important role in teaching, scientific research and medical examination.

Successful orthodontic treatment is based on a comprehensive diagnosis and treatment planning. A few of the fundamental factors in the diagnosis are the spacing condition, tooth size, arch form and dimensions, as well as the tooth-arch discrepancies. Intraoral photographs' major role is to enable orthodontists to document and analyze the occlusal relationships as well as the dental and soft-tissue features in order to arrive at a good diagnosis and an appropriate treatment plan.

In 1975, Robert Little developed Little's irregularity index (LII). The index was proposed to assess teeth irregularity, crowding, relapse, and alignment of anterior teeth as it measured the linear displacements in the horizontal plane between contact points of anterior teeth, ignoring vertical displacement, from mesial surface of one canine to the contra-lateral one. The sum of the 5 liner measurements of displacements was the LII score. The higher the index value, the more severe irregularity of the teeth was. LII has been originally developed for mandibular incisors to study relapse; however, researchers have used it to assess upper and lower incisors irregularity

Tooth-size-arch-length discrepancy (TSALD) is widely used on study models to assess the level of harmony between tooth size and the supporting basal bone. Bolton analysis is another important measurement used to identify disharmony between maxillary and mandibular tooth size which is considered an important factor to ensure the success of orthodontic treatment. With the application of the suggested formulas, the overall ratio should be 91.3% (±1.91) and the partial (anterior) ratio should be 77.2% (±1.65).

The validity and reliability of performing the above mentioned analyses on images taken of the dental arches have not been evaluated yet in the literature. This is the aim of the current project.

DETAILED DESCRIPTION:
Assessment of the LII scores, TSALD, Bolton analysis has been performed by the majority of previous studies using plaster models and calipers in a direct manner. Others have measured previous variables indirectly using 2-dimensional and 3-dimensional (3D) methods. 2D methods have included 2D scans of plaster models or 2D images of the occlusal views. The obtained images have been then analyzed either manually or on-screen using dedicated software. 3D methods have included digital models and have been used by several researchers. Although the wealth of knowledge 3D methods provide, they require the use of 3D imaging techniques with the resultant additional costs, time and labor.

Many studies have used 2D digital images of poured plaster models to perform software-based measurements of tooth movement during active treatment but these studies have not reported the accuracy and reproducibility of their methods. Dental impressions have been required to obtain proper study models. This procedure is a time- and labor-consuming for the orthodontist and could be exhausting to the patient. When braces are fitted, impression taking becomes a difficult task and if several impressions are required in the context of a research project, this would impose additional burden to patients and researchers. Therefore, taking intra-oral images of dental arches instead of impressions seems to be a very convenient alternative.

Validity and reliability of measurements made on photographs of study models have been evaluated in previous reports. However, it seems to be that there is only one paper in the literature with the aim of validating the use of intra-oral images of the dental arches for performing dental measurement. They found that the analysis of LII was valid. However, the practicability of their suggested method of imaging was questionable and their evaluation was only confined to the LII, which is not the only variable that is used in our ordinary plaster model analysis.

Therefore, the primary aim of the current work were to evaluate the validity and reliability of measurements made directly on intraoral photographs compared to those made on poured plaster models in the assessment of the LII, TSALD, and Bolton ratios. As a secondary aim, the comparisons were also accomplished with those measurements made on photographs taken of the corresponding poured plaster models .

ELIGIBILITY:
Inclusion Criteria:

* Complete permanent dentition
* Absence of any big carious lesions
* Absence of fixed prosthodontics (fixed bridges)
* Absence of shape and size disturbances (regardless third molar)
* Presence of upper and lower crowded arches

Exclusion Criteria: (fixed br

* Missing teeth
* Migrated teeth
* Impacted teeth
* Severely broken down teeth or big carious lesions
* Presence of fixed prosthodontics (fixed bridges)
* Presence of shape and size disturbances

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with different levels of malocclusion
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-08-19 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Little's Index of Irregularity (LII) | After seven days of taking the impressions of the dental arches. Impressions will be taken in the same day of patient's entry to the cohort.
  Robert Little developed Little's irregularity index (LII) in 1975. The index has been proposed to assess teeth irregularity, crowding, relapse, and alignment of anterior teeth as it measured the linear displacements in the horizontal plane between contact points of anterior teeth, ignoring vertical displacement, from mesial surface of one canine to the contra-lateral one. The sum of the 5 liner measurements of displacements is considered the LII score. The higher the index value, the more severe irregularity of the teeth is. LII has been originally developed for mandibular incisors to study relapse; however, researchers have used it to assess upper and lower incisors irregularity.
Partial Bolton's Ratio | After seven days of taking the impressions of the dental arches. Impressions will be taken in the same day of patient's entry to the cohort.
  Bolton analysis is used to identify disharmony between maxillary and mandibular tooth size which is considered an important factor to ensure the success of orthodontic treatment. With the application of the suggested formula, the partial ratio should be 77.2% (±1.65)
  The formula is the sum of the mesio-distal widths of the lower six anterior teeth divided by the sum of the mesio-distal widths of the upper six anterior teeth.
Overall Bolton's Ratio | After seven days of taking the impressions of the dental arches. Impressions will be taken in the same day of patient's entry to the cohort.
  Bolton analysis is used to identify disharmony between maxillary and mandibular tooth size which is considered an important factor to ensure the success of orthodontic treatment. With the application of the suggested formula, the overall ratio should be 91.3%.
  The formula is the sum of the mesio-distal widths of the lower twelve teeth divided by the sum of the mesio-distal widths of the upper twelve teeth.
Tooth-size-arch-length-discrepancy (TSALD) | After seven days of taking the impressions of the dental arches. Impressions will be taken in the same day of patient's entry to the cohort.
  Tooth-size-arch-length discrepancy (TSALD) is widely used on study models to assess the level of harmony between tooth size and the supporting basal bone.
  The formula is The sum of mesio-distal widths of all permanent teeth (mesial to the first lower/upper molars) minus the sum of the basal bone length (measured by a specific thread). The result is expressed in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Wael Al-Rasheed Omer, DDS, Principal Investigator — MSc student at the Orthodontic Department, University of Damascus Dental School, Damascus, Syria; Amer M Owayda, DDS, Principal Investigator — MSc student in Orthodontics, University of Damascus Dental School, Damascus, SYRIA; Mohammad Y Hajeer, DDS MSc PhD, Study Director — Associate Professor of Orthodontics, University of Damascus Dental School, Damascus, SYRIA; Rashad Murad, DDS MSc PhD, Study Director — Associate Professor of Toxicology, University of Damascus Pharmacological College, Damascus, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almasoud N, Bearn D. Little's irregularity index: photographic assessment vs study model assessment. Am J Orthod Dentofacial Orthop. 2010 Dec;138(6):787-94. doi: 10.1016/j.ajodo.2009.01.031. PMID 21130338
- [Background] Jones ML. The Barry Project--a three-dimensional assessment of occlusal treatment change in a consecutively referred sample: the incisors. Br J Orthod. 1990 Feb;17(1):1-19. doi: 10.1179/bjo.17.1.1. PMID 2310735
- [Background] Little RM. The irregularity index: a quantitative score of mandibular anterior alignment. Am J Orthod. 1975 Nov;68(5):554-63. doi: 10.1016/0002-9416(75)90086-x. PMID 1059332
- [Background] Puneky PJ, Sadowsky C, BeGole EA. Tooth morphology and lower incisor alignment many years after orthodontic therapy. Am J Orthod. 1984 Oct;86(4):299-305. doi: 10.1016/0002-9416(84)90140-4. PMID 6592978
- [Background] Surbeck BT, Artun J, Hawkins NR, Leroux B. Associations between initial, posttreatment, and postretention alignment of maxillary anterior teeth. Am J Orthod Dentofacial Orthop. 1998 Feb;113(2):186-95. doi: 10.1016/s0889-5406(98)70291-4. PMID 9484210
- [Background] Tran AM, Rugh JD, Chacon JA, Hatch JP. Reliability and validity of a computer-based Little irregularity index. Am J Orthod Dentofacial Orthop. 2003 Mar;123(3):349-51. doi: 10.1067/mod.2003.76. No abstract available. PMID 12637908
- [Background] West AE, Jones ML, Newcombe RG. Multiflex versus superelastic: a randomized clinical trial of the tooth alignment ability of initial arch wires. Am J Orthod Dentofacial Orthop. 1995 Nov;108(5):464-71. doi: 10.1016/s0889-5406(95)70046-3. PMID 7484965